CLINICAL TRIAL: NCT07146607
Title: Audiology Text-Messaging Intervention (Florence) to Improve Hearing Aid Use in NHS Adult Audiology Patients: A Feasibility Study With Proof-of-Concept and Embedded Process Evaluation
Brief Title: Evaluating an Audiology Text-Message Protocol to Support Hearing Aid Use in NHS Adult Audiology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WSAUD A/S (Industry)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Nottingham (Other)
Responsible Party: Principal Investigator, Emma Broome, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 345347
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aid; health behaviour
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing aids plus text-message protocol (Experimental): Audiology text-message protocol: The experimental group will receive a minimum of 65 text-messages directly to their mobile telephone for the duration of the 14-week text-message protocol (2 weeks for Stage 1 protocol, 12 weeks for Stage 2 protocol) in addition to receiving the standard audiology treatment as usual (see Control: Standard audiological care (hearing aid provision - treatment as usual)).
  Interventions: Behavioral: Audiology text-message protocol
- Standard audiological care (treatment as usual) (No Intervention): Participants allocated to the control group will receive treatment as usual. Treatment as usual is defined as standard treatment available to NHS audiology patients. This may include an audiological assessment, prescription of one/two hearing aids, and an optional face-to-face follow-up appointment.

INTERVENTIONS:
Behavioral: Audiology text-message protocol — Florence is an interactive text messaging service, endorsed by NHS England, designed to improve clinical outcomes for patients. An audiology text-message protocol, delivered via Florence, will prepare, inform and support new NHS hearing aid users as they are prescribed, receive, and start to use their hearing aid(s).
  Arms: Hearing aids plus text-message protocol

SUMMARY:
Over 18 million adults in the United Kingdom have significant hearing loss, linked to isolation, depression and comorbidities. Hearing aids are the main management option yet are frequently unused (~23%) or used irregularly (<40%), wasting NHS resources and reducing quality-of-life gains. Digital behaviour-change interventions can improve self-management between appointments. Florence, an NHS-endorsed text-messaging system, has been used in the management of other long-term conditions, but has not yet been applied within audiology. This study will test a standardised audiology text-message protocol, delivered via Florence, to support new NHS hearing aid users, aiming to improve adherence, outcomes, and cost-effectiveness. Outcomes assess trial feasibility (primary objective), proof-of concept for efficacy (secondary objective), and process evaluation (tertiary objective).

DETAILED DESCRIPTION:
Over 18 million adults in the UK have significant hearing loss, with prevalence and severity increasing with age. Hearing loss is a leading global cause of disability, associated with social isolation, depression, dementia, and reduced quality of life, and is more common among people with other long-term conditions such as diabetes, hypertension, and cardiovascular disease. Hearing aids are the standard clinical management, yet up to 23% of new users abandon them and <40% use them irregularly, resulting in wasted NHS resources and prolonging hearing difficulties.

Adjusting to hearing aids is a novel health behaviour, and behaviour-change interventions informed by health psychology can empower patients to manage their care, benefiting both patients and healthcare systems. Digital interventions, such as mobile text-messaging, are cost-effective ways to provide information and support between appointments and improve self-management.

Florence, an NHS-endorsed text-messaging system, has improved self-management in long-term conditions including hypertension, diabetes, and cancer, improving patient satisfaction and cost-effectiveness. It has not yet been applied in audiology. This feasibility study will examine a standardised audiology text-message protocol, delivered via Florence, for new NHS hearing aid users, addressing trial feasibility, proof-of-concept, and process evaluation objectives. Effective use could improve hearing aid adherence, quality of life, and save the NHS millions annually.

ELIGIBILITY:
WP1: Pilot Feasibility Study (n=60, 30 per group intervention/control (treatment as usual)) Inclusion criteria

* Aged ≥18 years (no upper age limit)
* Prescribed their first NHS acoustic hearing aid(s) for the primary concern of hearing loss
* Able and willing to provide informed consent
* Not currently participating in similar research
* Access to a mobile device (This is not required to be a smart phone device)

Exclusion criteria

* Registered on a pre-existing Florence text-messaging protocol.
* Unable to read/understand English

WP2: Nested Process Evaluation (minimum n=10 patients, n=2 clinicians) Inclusion criteria (patients)

* Aged ≥18 years (no upper age limit)
* Prescribed their first NHS acoustic hearing aid(s) for the primary concern of hearing loss
* Able and willing to provide informed consent

Exclusion criteria (patients)

* Registered on a pre-existing Florence text-messaging protocol.
* Unable to read/understand English

Inclusion criteria (clinicians)

* Aged ≥18 years (no upper age limit)
* Able and willing to provide informed consent

Exclusion criteria (clinicians)

• Not meeting criteria for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported hearing aid use | From enrollment to week 16 and 28
  A bespoke single item question recording the self-reported average hours of daily hearing aid use over the past seven days. The question "On a typical day over the last seven days, how many hours did you use your hearing aid?" will be collected via participants' preferred contact method.
Glasgow Hearing Aid Benefit Profile (GHABP): (Gatehouse 1999) | Week 1 (Part A) Week 16, 28 (Part B)
  The GHABP is a 24-item scale consisting of six subscales. The subscales address hearing aid initial disability, hearing aid handicap, reported hearing aid use, reported hearing aid benefit, hearing aid satisfaction and hearing aid derived benefit. Each domain is measured on a five-point scale, and the mean score across four predefined situations is converted into a percentage. Participants will only be asked to complete Part A (preintervention) of the GHABP questionnaire at the baseline assessment (pre-hearing aid fitting). Part B (residual) will be completed at the 16 and 28 week follow up (post-hearing aid fitting).

SECONDARY OUTCOMES:
Hearing Handicap Inventory for the Elderly/Adults (HHIE/A): (Ventry and Weinstein 1982) | Week 1, Week 16, 28
  The HHIE is a 25-item questionnaire designed to assess the effects of hearing loss on the emotional (n = 13), social and situational adjustment (n = 12) of older people, scored using a three-point scale (4 = yes; 2 = sometimes; 0 = no). A higher score indicates a more severe level of handicap.
Auditory Lifestyle and Demand questionnaire (ALDQ): (Gatehouse 1999) | Week 1, Week 16, 28
  The ALDQ (Gatehouse, 1999) is a questionnaire assessing auditory lifestyle. It describes a range of listening environments that are experienced by the PHL and the extent to which auditory requirements play a role in daily functioning. It is a 24-item questionnaire with two subscales: lifestyle and demand. Lifestyle scores are computed by totalling the 24 item responses in the subscale (maximum points 48). The demand subscale is calculated by multiplying the Lifestyle subscale with its corresponding importance weighting. The 24 products are then totalled to create a Demand score for the subject (maximum 96 points). Both the 'lifestyle' and 'demand' subscales are converted to percentage scores.
International Outcome Inventory for Hearing Aids (IOI-HA) (Cox and Alexander 2002) | Week 16, 28
  The IOI-HA consists of seven questions each probing a separate area related to hearing aid use including usage benefit, satisfaction, quality of life, impact on others and residual difficulties. Responses to the items are assigned a value of 1 to 5, with higher scores indicating a more favourable outcome.
Hearing Related Lifestyle (HEARLI-Q) (Lelic, Wolters et al. 2022) | Week 16, 28 Week 1, Week 16, 28
  The HEARLI-Q is a questionnaire consisting of 23 listening situations that participants rate on frequency of occurrence, importance to hear well, difficulty to hear and hearing aid satisfaction. Scores are calculated as follows:
  * Richness of Hearing-Related Lifestyle = (sum of all occurrence scores/92) × 100 in order to arrive at a score between 0 and 100.
  * Hearing Demand = (sum of [occurrence × importance]/368) × 100 in order to arrive at a score between 0 and 100.
  * Hearing Difficulty = average of the difficulty scores
  * Hearing Aid Satisfaction = average of the satisfaction scores excluding the response "I don't wear hearing aids in this situation." The situations in which participants do not wear hearing aids are reported alongside the overall hearing aids satisfaction score.
Hearing related adaptive strategies (AStra) (Fischer 2024) | Week 1, Week 16, 28
  The AStra questionnaire is an 18-item questionnaire assessing the type of strategies patients use in their everyday life to cope with hearing difficulties. Each item is rated on a seven-point scale ranging from never to always. Items are scores on three scales: i) selection; ii) optimization, iii) compensation. To score scale selection items 5 and 6 are inverted and the mean of items 1-6 is calculated. For scale optimisation the mean of items 7-12 is calculated and for scale compensation the mean of items 13-18 is calculated.
Big Five Inventory (BFI) (John 1991) | Week 1
  The BFI is a 44-item inventory that measures an individual on the Big Five Factors (dimensions) of personality. It comprised of five dimensions: i) extraversion versus introversion, ii) agreeableness versus antagonism, iii) conscientiousness versus lack of direction, iv) neuroticism versus emotional stability, v) openness versus closedness to experience. Each item is rated on a five-point scale ranging from 1 (disagree strongly) to 5 (agree strongly). The following items should be reverse scores: Extraversion: items 6R, 21R, 31R; Agreeableness: items 2R, 12R, 27R, 37R; Conscientiousness: items 8R, 18R, 23R, 43R; Neuroticism: items 9R, 24R, 34R; Openness: items 35R, 41R. After reverse scoring, find the total score for E(Extroversion), A (Agreeableness), C (Conscientiousness), N (Neuroticism), and O (Openness).
Short Assessment of Patient Satisfaction (SAPS) (Hawthorne, Sansoni et al. 2014) | Week 1, 28
  A seven-item scale that assesses patient satisfaction with their treatment. It assesses the core domains of patient satisfaction which include treatment satisfaction, explanation of treatment results, clinician care, participation in medical decision making, respect by the clinician, time with the clinician, and satisfaction with hospital/clinic care. Responses scales are on a 5-point scale. To score, reverse the scores for items 1, 3, 5 and 7; then sum all scores. The score range is from 0 (extremely dissatisfied) to 28 (extremely satisfied).
Measure of Audiologic Rehabilitation Self-Efficacy for Hearing Aids (MARS-HA): (West and Smith 2007) | Week 1, Week 16, 28
  The MARS-HA is a 24 item self-assessment of a patient's ability to do certain activities with a hearing aid as well as the patient's abilities to hear in certain situations. The MARS-HA measures four factors: 1) Basic Handling, 2) Advanced Handling, 3) Adjustment, and 4) Aided Listening. The MARS-HA subscale and total scale scores are calculated by taking the average of the item responses. An average less than or equal to 80% indicates a low or moderate self-efficacy.
Short Form Patient Activation Measure (PAM) (Hibbard, Mahoney et al. 2005) | Week 1, 3, 16, 28
  A 13-item validated questionnaire assesses the knowledge, skills, and confidence of patients to self-manage their health. Participants indicated how much each statement applies to them on a four-point scale: 0 (disagree strongly) to 3 (agree strongly). Scores are summed and converted into an activation score between 0-100 (0 = no activation, 100 = high activation).
Empowerment Audiology Questionnaire (EmpAQ-15) (Bennett, Larsson et al. 2024) | Week 1, 3, 16, 28
  the EmpAQ -15 is a 15 item questionnaire to measure empowerment in adults with hearing loss. Participants respond to items using a 4 point Likert scale ranging from strongly disagree to strongly agree. Each item is scored on a scale from 1 to 4 (e.g. strongly disagree = 1). Not applicable is scored as missing. Calculate the mean score by summing the response scores divided by the number of items answered. Subtract 1 and multiply by 33.33. The final score is presented as a scale with a range between 0-100% with a high % indicating a higher level of empowerment.
Expected Consequences of Hearing aid Ownership (ECHO): (Cox and Alexander 2000) | Week 1, 3, 16, 28
  The ECHO is a 15-item questionnaire for measuring expectations about hearing aids. There are four subscales: positive effect, service and cost, negative features and personal image. The response to each item is scored from 1-7. For all subscales, a higher score is indicative of a more favourable inclination toward the hearing aid. In the 'negative features' subscale, a higher score can be interpreted as reflecting a lack of knowledge or concern about potentially problematic issues. An average score is calculated for each subscale. The Global Score is the mean of the scores for all the items.
Stigma Consciousness Questionnaire for Hearing Loss (SCQ-HL): (Vincent, Gagné et al. 2017) | Week 1, 16, 28
  The SCQ-HL is a 10-item self-report questionnaire that measures the extent to which respondents expect to be stereotyped because of their disability, social role or sexual orientation. Each statement is rated on a seven-point scale ranging from 0 (completely disagree) to 6 (completely agree). The scale includes a midpoint of 3, denoting 'neither agree nor disagree'. A high total score indicates that a respondent's level of stigma consciousness is high.
Patient Global Impression Scale - Improvement (PGI-I) (Guy, 1976) | Week 16, 28
  The PGI-I is a one-item questionnaire that asks an individual patient to rate at endpoint the perceived change in his/her daily listening and communication in response to an intervention. It is rated on a seven-point scale ranging from 1 (very much better) to 7 (very much worse). A low score indicates that respondent's daily listening and communication is very much better than before wearing hearing aids.
Health Utilities Index (HUI-III) (Feeny, Furlong et al. 2002) | Week 1, 16, 28
  The HUI-III measures health-related quality of life. It comprises of eight attributes (Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition and Pain) within each attribute there are five or six levels of ability/disability.
EQ-5D-3L (Oppe, Devlin et al. 2014) | Week 1, 16, 28
  The EQ -5D-3L comprise of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The patient indicates their health status by ticking the box next to the most appropriate statement in each dimension ranging from no problems to extreme problems. Each health state can be assigned a summary index score ranging from 0 to 1, with higher scores indicating high health utility.
Data logging from the text-message intervention | Week 28
  Data such as text-message receipt data, how many reminder messages were sent and the number of participants who opted-out of the text-messages will be recorded directly from the Florence telehealth system. Other information such as the type of goals/plans set within the text-message intervention and patient keyword text inputs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Emma E Broome, PhD, Principal Investigator — University of Nottingham
Locations (1):
- QMC Ropewalk House, Nottingham, Nottinghamshire, United Kingdom